CLINICAL TRIAL: NCT06703645
Title: Evaluation of Snakebite Cases in Assiut Governorate, Egypt (Prospective Study)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Alkady Mohamed, Demonstrator, Assiut University
Other Study IDs: Snakebites in Assiut Governate
Record Dates: First submitted 2024-11-17; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Snakebite Cases Evaluation Clinical and Laboratory
Keywords: snakebite
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. Study the sociodemographic profile of snakebite victims in Assiut Governorate.
2. Portray the clinical profile of snakebite victims admitted to Assiut University , El Eman General Hospital and Assiut General Hospital.
3. Assess the predictors of severity and outcome of cases.

DETAILED DESCRIPTION:
Snake's envenomation is a serious socio-medical problem, which causes considerable mortality and morbidity, with approximately 125,000 deaths worldwide annually. There were 4.5 to 5.4 million bites every year, and of those figures, 40-50% had some clinical disability as a result. Furthermore, the death from such an issue could go somewhere between 80,000 and 130,000 individuals each year. In the Middle East and North Africa, there are over 70,000 snakebites bites each year.

There are many species of snakes, approximately 3,700 species of snakes worldwide only about 15% are venomous belong to the four large families including Viperidae, Colubridae, Elapidae and Atractaspidinae. Two of these toxic species are widespread in Egypt; the family Viperidae and the family Elapidae Egyptian copra Naja Haje.

Snake venoms are complex mixtures consisting of enzymatic components e.g., proteolytic enzymes e.g., serine protease and metalloproteases (SVMPs), non-enzymatic components e.g., cysteine-rich secretory proteins (CRISP), amines, lipids, nucleotides, and carbohydrates. Venoms also contain inorganic cations that are presumed to function as cofactors and include sodium, calcium, potassium, magnesium, and zinc.

Snake venoms are usually classified as hemotoxic or neurotoxic. Snakes of the Viperidae family have venom containing proteins that can disrupt the coagulation cascade, the hemostatic system and tissue integrity. In contrast, neurotoxic venoms, which are typical of the Elapidae snakes, contain several toxins that primarily affect the peripheral nervous system, in particular the neuromuscular junction.

Depending on the species of snakes, manifestations can be localized symptoms of mild pain, progressive edema, ecchymosis, and tissue necrosis and generalized ones as spontaneous bleeding e.g., bleeding per gums, epistaxis, hematuria, vaginal bleeding, hematemesis, hematochezia, hemoptysis, hemolytic anemia and hemolytic jaundice with hemototoxic snake venom. In severe cases patients may develop acute renal, myocardial infarction, disseminated intravascular coagulation, or even death. Ptosis, diplopia, dysphagia, trunk and limbs weakness, and respiratory paralysis which can lead to respiratory failure and apnea with neurotoxic snake venom.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with a reliable history of snakebite.
* Presence of fang marks and/or signs of local and systemic envenomation.

Exclusion Criteria:

* Fake or uncertain snakebites.
* Patients with history of hematological disorders, liver diseases, renal diseases and anticoagulation therapy in the past week.
* Patients who are not willing to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases will be collected from emergency departments, inpatient units of Assiut University Hospitals, El Eman General Hospital and Assiut General Hospital. All cases will be evaluated by detailed history, examination, investigations and through sheet which consist of:
  1. Detailed information regarding demographic and epidemiological parameters such as age, sex, residence, occupation, site, time and place of bite in addition to type of snake if identification was obtained.
  2. Clinical manifestations:
     * Local manifestations
     * Systemic manifestations
       * Hematological e.g., spontaneous bleeding like epistaxis, hematemesis, melena, and hematuria.
       * Neurological e.g., ptosis, dysphonia, dysphagia, and descending paralysis.
       * Cardiovascular e.g., dizziness, palpitation, faintness, hypotension, cardiac arrhythmias, and shock.
       * Respiratory e.g., tachypnea and shortness of breathing
     * The severity of envenomation will be assessed using the scoring and grading systems
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with recovery | through study completion, an average of 1 year".
  1. Number of Participants with complete recovery.
  2. Number of Participants with recovery with disability and complications as amputation and renal failure, etc.
Number of Participants with Death | through study completion, an average of 1 year".
  Any complication due to snake bite end with death as respiratory arrest, disseminated intravascular coagulation and renal failure.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohammed Fathy, Professor, Study Director — Assiut University; Nora Zeidan Abdellah, Assistant lecture, Study Director — Assiut University

REFERENCES:
- [Background] Padhiyar R, Chavan S, Dhampalwar S, Trivedi T, Moulick N. Snake Bite Envenomation in a Tertiary Care Centre. J Assoc Physicians India. 2018 Mar;66(3):55-9. PMID 30341870
- [Background] Namal Rathnayaka R, Ranathunga PAN, Kularatne SA. Thrombotic Microangiopathy, Hemolytic Uremic Syndrome, and Thrombotic Thrombocytopenic Purpura Following Hump-nosed Pit Viper (Genus: Hypnale) Envenoming in Sri Lanka. Wilderness Environ Med. 2019 Mar;30(1):66-78. doi: 10.1016/j.wem.2018.10.003. Epub 2019 Jan 31. PMID 30711421
- [Background] Langley R, Haskell MG, Hareza D, King K. Fatal and Nonfatal Snakebite Injuries Reported in the United States. South Med J. 2020 Oct;113(10):514-519. doi: 10.14423/SMJ.0000000000001156. PMID 33005969
- [Background] Kumar KS, Narayanan S, Udayabhaskaran V, Thulaseedharan NK. Clinical and epidemiologic profile and predictors of outcome of poisonous snake bites - an analysis of 1,500 cases from a tertiary care center in Malabar, North Kerala, India. Int J Gen Med. 2018 Jun 5;11:209-216. doi: 10.2147/IJGM.S136153. eCollection 2018. PMID 29892202
- [Background] Kang S, Moon J, Chun B. Does the traditional snakebite severity score correctly classify envenomated patients? Clin Exp Emerg Med. 2016 Mar 31;3(1):34-40. doi: 10.15441/ceem.16.123. eCollection 2016 Mar. PMID 27752613
- [Background] Jenkins TP, Ahmadi S, Bittenbinder MA, Stewart TK, Akgun DE, Hale M, Nasrabadi NN, Wolff DS, Vonk FJ, Kool J, Laustsen AH. Terrestrial venomous animals, the envenomings they cause, and treatment perspectives in the Middle East and North Africa. PLoS Negl Trop Dis. 2021 Dec 2;15(12):e0009880. doi: 10.1371/journal.pntd.0009880. eCollection 2021 Dec. PMID 34855751
- [Background] Isbister GK. Snakebite doesn't cause disseminated intravascular coagulation: coagulopathy and thrombotic microangiopathy in snake envenoming. Semin Thromb Hemost. 2010 Jun;36(4):444-51. doi: 10.1055/s-0030-1254053. Epub 2010 Jul 7. PMID 20614396
- [Background] Harris JB, Scott-Davey T. Secreted phospholipases A2 of snake venoms: effects on the peripheral neuromuscular system with comments on the role of phospholipases A2 in disorders of the CNS and their uses in industry. Toxins (Basel). 2013 Dec 17;5(12):2533-71. doi: 10.3390/toxins5122533. PMID 24351716
- [Background] Bickler PE. Amplification of Snake Venom Toxicity by Endogenous Signaling Pathways. Toxins (Basel). 2020 Jan 22;12(2):68. doi: 10.3390/toxins12020068. PMID 31979014